CLINICAL TRIAL: NCT02417454
Title: A Double Blind Placebo Controlled Study on the Effects of a Probiotic on Autonomic and Psychological Stress Responses in Volunteers
Brief Title: Study on the Effects of a Probiotic on Autonomic and Psychological Stress
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Lallemand Health Solutions (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20000229
Record Dates: First submitted 2015-04-07; First posted 2015-04-15 (Estimated); Last update posted 2017-10-19 (Actual); Status verified 2017-10

CONDITIONS: Stress, Psychological
Keywords: probiotic; stress; emotion psychophysiology; brain-body-gut interactions
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Probiotic (Experimental): Participants will undergo the same study procedures as for the comparator; however, the product given will be the active probiotic supplement (ProbioStick).
  Interventions: Dietary Supplement: ProbioStick
- Placebo (Placebo Comparator): Participants will undergo the same study procedures as for the probiotic; however, the product given will be a placebo, identical to the probiotic in taste, smell, colour, and comprised only of the same non-active ingredients in the probiotic supplement
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: ProbioStick — One sachet daily, without or without meals (3 x 10^9 CFU per sachet)
  (Lactobacillus helveticus R0052 and Bifidobacterium longum subsp. longum R0175)
  Arms: Probiotic
Other: Placebo — One sachet daily, without or without meals (0 CFU per sachet)
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the effects of a probiotic blend on qualitative (subjective interviews and self-reporting) and quantitative (changes in brain activity, heart rate, cortisol, and reactivity) measures of stress in healthy undergraduate students.

DETAILED DESCRIPTION:
There is a burgeoning literature involving nonhuman animal and human studies linking the microbiota environment in the gut to brain-behaviour relations. For example, animal studies demonstrate that germ-free rodents show heightened HPA-axis responses to stress compared to gnotobiotic animals. There are also a number of nonhuman and human studies that show positive effects of reducing stress after being treated with different probiotics. For example, in one recent double blind study in humans using standardized questionnaires indicated a greater reduction of stress and anxiety symptoms after one month of supplementation with a probiotic formulation compared to placebo. The groups were also differentiated by urinary cortisol levels after treatment. Other studies have found positive effects of probiotic treatment and stress reduction using other probiotics. Accordingly, there is accumulating empirical evidence from animal and human studies of the positive effects of probiotic treatment on stress reduction.

In this study, the investigators will investigate the stress reduction effects of the Lallemand Health Solutions (LHS) Probio'Stick® on healthy undergraduate students. The study will be conducted at the McMaster LIVELab, which is capable of collecting both physiological and behavioural measures from groups of up to 100 participants at a time.

Registration into this clinical trial will require students be screened via McMaster's SONA system (mcmaster.sona-systems.com). After the screening, participants that are eligible to participate will be given the option to register for an information meeting at which point one may opt to enrol in the study or not.

Once in the study, participants will undergo an initial screening in the LIVELab where they will be exposed to auditory, visual, and performance based stressors to measure a baseline. After such point, they will be randomized to receive Probio'Stick® or placebo for a 6-week, once daily, probiotic treatment at home. Following the 6 week intervention, participants will return to the lab for a second testing using the same procedures to establish a change from baseline.

ELIGIBILITY:
Inclusion Criteria:

* Answering "Yes" to questions 3, 8 and 9 of the Cohen's Perceived Stress Scale.
* Willingness to complete questionnaires, records, and diaries associated with the study and to complete all site visits.
* Willingness to discontinue consumption of fermented foods or probiotics (e.g. yogurts, with live, active cultures, or supplements).
* Ability to provide informed consent.

Exclusion Criteria:

* Must not be currently taking another probiotic regiment or another investigational product within 3 months of the screening visit.
* Must not currently be taking medications for depression or anxiety, including benzodiazepines, SSRIs, or antipsychotics or receiving counselling for depression or anxiety.
* Must not be immune-compromised or immuno-suppressed (e.g. AIDS, lymphoma, participants undergoing long-term corticosteroid treatment, chemotherapy and allograft participants).
* Must not have experienced bloody diarrhea in the past month prior to beginning the study.
* Must not have undergone any surgery within the three months prior to beginning the study, particularly surgeries involving the colon.
* Must not have any soy or milk allergy.
* Must not be pregnant or breast-feeding or planning on becoming pregnant.
* Must not have used of any antibiotic drug (e.g., neomycin, rifaximin) within 1 month of screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2015-09; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Changes in right frontal electroencephalography (EEG)/brain activity | Visit 1 and Visit 2 (6 weeks apart)
  Is a measure of stress/arousal
Changes in salivary cortisol concentrations | Pre and Post Visit 1 and Visit 2 (6 weeks apart)
  Collected via Salivette®, before and after each session in the lab.
Change in the magnitude of startle response | Visit 1 and Visit 2 (6 weeks apart)
  Measured as facial electromyography (EMG) change
Changes in sympathetic nervous system activation | Visit 1 and Visit 2 (6 weeks apart)
  Calculated as a measure of Heart Rate Variability (HRV) from electrocardiography (ECG) data

SECONDARY OUTCOMES:
Changes in Anxiety Scores as determined by the Beck Anxiety Inventory (BAI) | Visit 1 and Visit 2 (6 weeks apart)
Changes in Stress Scores as determined by Cohen's Perceived Stress Scale (PSS) | Visit 1 and Visit 2 (6 weeks apart)
Changes in General Affect Scores as determined by the Positive and Negative Affect Scale (PANAS) | Visit 1 and Visit 2 (6 weeks apart)
Changes in Stress Scores as reported on a 1-10 Likert Scale | Visit 1 and Visit 2 (6 weeks apart)

CONTACTS AND LOCATIONS:
Overall Officials: Laurel Trainor, Ph.D., Principal Investigator — McMaster University
Locations (1):
- McMaster LIVELab, Hamilton, Ontario, Canada

REFERENCES:
- [Background] Lutgendorff F, Akkermans LM, Soderholm JD. The role of microbiota and probiotics in stress-induced gastro-intestinal damage. Curr Mol Med. 2008 Jun;8(4):282-98. doi: 10.2174/156652408784533779. PMID 18537636
- [Background] Ait-Belgnaoui A, Colom A, Braniste V, Ramalho L, Marrot A, Cartier C, Houdeau E, Theodorou V, Tompkins T. Probiotic gut effect prevents the chronic psychological stress-induced brain activity abnormality in mice. Neurogastroenterol Motil. 2014 Apr;26(4):510-20. doi: 10.1111/nmo.12295. Epub 2013 Dec 30. PMID 24372793
- [Background] Ait-Belgnaoui A, Durand H, Cartier C, Chaumaz G, Eutamene H, Ferrier L, Houdeau E, Fioramonti J, Bueno L, Theodorou V. Prevention of gut leakiness by a probiotic treatment leads to attenuated HPA response to an acute psychological stress in rats. Psychoneuroendocrinology. 2012 Nov;37(11):1885-95. doi: 10.1016/j.psyneuen.2012.03.024. Epub 2012 Apr 26. PMID 22541937
- [Background] Palomar MM, Maldonado Galdeano C, Perdigon G. Influence of a probiotic lactobacillus strain on the intestinal ecosystem in a stress model mouse. Brain Behav Immun. 2014 Jan;35:77-85. doi: 10.1016/j.bbi.2013.08.015. Epub 2013 Sep 7. PMID 24016865
- [Background] Kullisaar T, Songisepp E, Mikelsaar M, Zilmer K, Vihalemm T, Zilmer M. Antioxidative probiotic fermented goats' milk decreases oxidative stress-mediated atherogenicity in human subjects. Br J Nutr. 2003 Aug;90(2):449-56. doi: 10.1079/bjn2003896. PMID 12908907
- [Background] Messaoudi M, Violle N, Bisson JF, Desor D, Javelot H, Rougeot C. Beneficial psychological effects of a probiotic formulation (Lactobacillus helveticus R0052 and Bifidobacterium longum R0175) in healthy human volunteers. Gut Microbes. 2011 Jul-Aug;2(4):256-61. doi: 10.4161/gmic.2.4.16108. Epub 2011 Jul 1. No abstract available. PMID 21983070
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Lang PJ, Bradley MM, Cuthbert BN. International affective picture system (IAPS): Affective ratings of pictures and instruction manual.. Technical Report A-8. University of Florida, Gainesville, FL.; 1995.
- [Background] Gasser F. Safety of lactic acid bacteria and their occurrence in human clinical infections. Bull Inst Past. 1994;92:45-67.
- [Background] Salminen S, von Wright A, Morelli L, Marteau P, Brassart D, de Vos WM, Fonden R, Saxelin M, Collins K, Mogensen G, Birkeland SE, Mattila-Sandholm T. Demonstration of safety of probiotics -- a review. Int J Food Microbiol. 1998 Oct 20;44(1-2):93-106. doi: 10.1016/s0168-1605(98)00128-7. PMID 9849787
- [Background] European Food Safety Authority (EFSA). Technical guidance - Update of the criteria used in the assessment of bacterial resistance to antibiotics of human or veterinary importance. EFSA J. 2008 Jul 14;6(7):732. doi: 10.2903/j.efsa.2008.732. eCollection 2008 Jul. No abstract available. PMID 37213835
- [Background] Garneau P, Labrecque O, Maynard C, Messier S, Masson L, Archambault M, Harel J. Use of a bacterial antimicrobial resistance gene microarray for the identification of resistant Staphylococcus aureus. Zoonoses Public Health. 2010 Nov;57 Suppl 1:94-9. doi: 10.1111/j.1863-2378.2010.01358.x. PMID 21083822
- See also: McMaster LIVELab — http://livelab.mcmaster.ca
- See also: McMaster SONA Recruitment — http://mcmaster.sona-systems.com